CLINICAL TRIAL: NCT04137861
Title: Evaluation of Furcal Perforation Repair in Primary Molars With MTA Versus Bioceramics
Brief Title: Evaluation of Furcal Perforation Repair in Primary Molars With MTA Versus Bioceramics (A Randomized Clinical Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmad Elheeny (Other)
Responsible Party: Sponsor-Investigator, Ahmad Elheeny, Clinical Professor, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 308
Record Dates: First submitted 2019-10-20; First posted 2019-10-24 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Iatrogenic Perforation of Primary Molars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mineral Trioxide Aggregate (MTA) (Active Comparator): Root repair material
  Interventions: Other: Bioceramics
- bioceramics (Experimental): Root repair material
  Interventions: Other: Bioceramics

INTERVENTIONS:
Other: Bioceramics — root repair material

SUMMARY:
Furcal perforation is one of the most challenging procedural accidents during pulpotomy of primary molars and should be sealed as soon as possible to prevent bacterial invasion at perforation site and subsequent tooth extraction. The aim of the study is to compare bioceramics versus MTA as root repair material for treatment of furcal perforation in primary molars

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy children aged from 4 to 7 years
* No history of spontaneous pain or swelling
* No signs or symptoms of irreversible pulpits or loss of vitality
* Absence of radicular or priapical lesions.
* Accidental furcal perforation should be immediate or mediate (within two weeks) perforation in primary molars.

Exclusion Criteria:

* Children with systemic disease
* Presence of priapical lesions

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
clinical success | 9 months
  Visual oral examination
radiographic success | 9 months
  Radiolucency assessment (+/-)

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Egypt

REFERENCES:
- [Derived] Abdelmotelb MA, Gomaa YF, Khattab NMA, Elheeny AAH. Premixed bioceramics versus mineral trioxide aggregate in furcal perforation repair of primary molars: in vitro and in vivo study. Clin Oral Investig. 2021 Aug;25(8):4915-4925. doi: 10.1007/s00784-021-03800-3. Epub 2021 Jan 22. PMID 33483869